CLINICAL TRIAL: NCT01288703
Title: Computerized-Adaptive Testing: Feasibility In Women With Pelvic Floor Disorders
Brief Title: Computerized-Adaptive Testing: Feasibility In Women With Pelvic Floor Disorders (CAT)
Acronym: CAT
Status: Completed | Type: Observational
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Vivian Sung, Principal Investigator, Women and Infants Hospital of Rhode Island
Other Study IDs: 10-0050
Record Dates: First submitted 2011-01-28; First posted 2011-02-02 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this pilot-study is to evaluate the feasibility and acceptability of PROMIS computerized-adaptive testing in women with urinary incontinence.

DETAILED DESCRIPTION:
Patient-reported outcomes (PRO's) are important to assess treatment progress in the field of pelvic floor disorders (PFDs), including urinary incontinence, pelvic organ prolapse, and fecal incontinence. The NIH has invested in the Patient-Reported Outcomes Measurement System (PROMIS) to revolutionize PRO measures. To date, PROMIS instruments and feasibility and acceptability of PROMIS and Computerized-Adaptive Testing (CAT) technology has not been well explored in women with PFDs and warrant further investigation. In recruiting sixty women, the investigators will conduct pilot-testing on the CAT mode of the PROMIS questionnaires, and compare participant's attitudes about the paper short-forms versus the CAT modes of administration.

The investigators will recruit 60 women with UI to participate in this study. Participants will be asked to complete both paper and CAT versions of PROMIS questionnaires covering the physical, social and mental health domains (Appendix 1). The time it takes to complete each version will be recorded. After completing the questionnaires, all participants will be interviewed, which will include a brief "Usability and Satisfaction Questionnaire"(Appendix 2), questions about technical problems, preferences, and the acceptability of each mode.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Able to read English
* Diagnosis of urinary incontinence
* Age 18 or older

Exclusion Criteria:

* Unable to read English or cognitive limitations making it difficult for study participants to complete PROMIS questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 women seeking care for PFDs will be eligible. Women will be excluded if they are unable to read English or have cognitive limitations precluding the completion of PROMIS questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 1 day
  To test the feasibility and acceptability of PROMIS and Computerized-Adaptive Testing (CAT) technology in women with Urinary incontinence. In recruiting sixty women, we will conduct pilot-testing on the CAT mode of the PROMIS questionnaires, and compare participant's attitudes about the paper short-forms versus the CAT modes of administration.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian W Sung, MD, MPH, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital Division of Urogynecology, Providence, Rhode Island, United States

REFERENCES:
- [Result] Sung VW, Marques F, Rogers RR, Williams DA, Myers DL, Clark MA. Content validation of the patient-reported outcomes measurement information system (PROMIS) framework in women with urinary incontinence. Neurourol Urodyn. 2011 Apr;30(4):503-9. doi: 10.1002/nau.21048. Epub 2011 Mar 11. PMID 21400574